CLINICAL TRIAL: NCT05147259
Title: A Single Center, Randomized, Double-Blind, Single Ascending Dose, Crossover Designed Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HR011408 at Two Formulations in Healthy Subject
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HR011408 at Two Formulations in Healthy Subject
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HR011408-101
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Diabetes in Adults

STUDY DESIGN:
Intervention Model Description: Crossover Assigned to HR011408(formulation A) or HR011408(formulation B)
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort one: Low dose (Experimental): Subjects will be randomized to a treatment sequence consisting of two treatment periods: received two formulation HR011408 injections successively
  Interventions: Drug: HR011408 injection
- Cohort two: Medium dose (Experimental): Subjects will be randomized to a treatment sequence consisting of two treatment periods: received two formulation HR011408 injections successively
  Interventions: Drug: HR011408 injection
- Cohort three: high dose (Experimental): Subjects will be randomized to a treatment sequence consisting of two treatment periods: received two formulation HR011408 injections successively
  Interventions: Drug: HR011408 injection

INTERVENTIONS:
Drug: HR011408 injection — Drug: HR011408 injection (formulation A), administered subcutaneously. Drug: HR011408 injection (formulation B), administered subcutaneously.

SUMMARY:
The objective of the study is to assess the safety, tolerability and pharmacokinetics of HR011408 at two formulations in healthy subject.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-55 years(both inclusive) at the time of signing informed consent
2. Body mass index 18.0-26.0kg/m2(both inclusive)
3. Body weight ≥50.0kg(male),≥45.0kg(female)
4. Fasting serum/plasma glucose <6.1mmol/L

Exclusion Criteria:

1. Known or suspected of being allergic to any ingredient in the study drug.
2. Participated in any drug or medical device-related clinical trial within 3 months before screening.
3. Subjects addicted to smoking, or non-smoker who smoked within 48 hours before administration
4. Donated blood within 1 month before screening; or donated blood ≥400 mL or had blood loss ≥400 mL during trauma or major surgery within 3 months before screening.
5. Subjects with incompetence or language impairment, who cannot fully understand or participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-02-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | from Day1 to Day15
  The incidence of adverse events will be collected and the safety of HR011408 will be assessed
Area under the concentration-time curve (AUC) | from 0 to 10 hours after dose administration
  Area under the concentration-time curve (AUC)
Maximum observed concentration (Cmax) | from 0 to 10 hours after dose administration
  Maximum observed concentration (Cmax)
Time to maximum observed concentration (Tmax) | from 0 to 10 hours after dose administration
  Time to maximum observed concentration (Tmax)
Elimination half-life (t1/2) | from 0 to 10 hours after dose administration
  Elimination half-life (t1/2)
Time to 50% maximum observed concentration (time to 50% Cmax) | from 0 to 10 hours after dose administration
  Time to 50% maximum observed concentration (time to 50% Cmax)
Onset of appearance | from 0 to 10 hours after dose administration
  First time point after dose administration when concentration reaches lower limit of quantification (LLOQ)

SECONDARY OUTCOMES:
Assessment of development of Anti-drug Antibodies (ADAs) | from Day1 to Day15 after dose administration
  Incidence of Anti-drug Antibodies (ADAs) will be assessed

IPD SHARING:
Plan to Share IPD: Undecided